CLINICAL TRIAL: NCT05543876
Title: The Effect of Video Watching With Virtual Reality Glasses on Pain and Fear of Children Presenting to the Emergency Department for Suture: A Randomized Controlled Study
Brief Title: The Effect of Video Watching With Virtual Reality Glasses on Pain and Fear of Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zühal Artuvan (Other)
Responsible Party: Sponsor-Investigator, Zühal Artuvan, Specialist Nurse, Mersin University
Organization: Mersin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Zühal Artuvan
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Child; Pain; Fear; Suture; Virtual Reality
Keywords: suture; virtual reality glasses; pain; fear; child
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): group watching video with virtual reality glasses
  Interventions: Procedure: suturing procedure
- control group (No Intervention): without any intervention

INTERVENTIONS:
Procedure: suturing procedure — Children presenting to the emergency department for suturing
  Arms: intervention group

SUMMARY:
IInvasive procedures such as suturing cause pain and fear in children. The high level of pain and fear of children makes it difficult to adapt to the procedure. It is a randomized controlled study planned to examine the effect of watching videos with virtual reality glasses as a distraction method while suturing in 7-12 age group children. Araştırma Acil Müdahale Odasında 01 Ekim 2022-31 Mart 2023 tarihlerinde yürütülmesi planlanmaktadır. In the collection of data; It is planned to use the Child Information Form, Wong-Baker Pain Scale, Child Fear Scale, which was created as a result of the literature review.

DETAILED DESCRIPTION:
TChildren may feel pain and fear during invasive procedures in the emergency room. The methodology of the research planned to be conducted in the Emergency Service with the participation of 84 children who met the inclusion and exclusion criteria between 01 October 2022 and 31 March 2023 is explained below. Children who apply to the emergency department due to an incision come to the emergency room and suturing takes place in this room. Two nurses work in this room, which is approximately 20 square meters, located at the entrance of the emergency room. G*Power 3.1.9.4 program was used to determine the number of children to be included in the study and control groups. In order for the difference between the study and control groups to be statistically significant in the study to be conducted, taking into account the previous studies, a total of at least 84 children (42 studies, 42 control groups) with 0.55 effect size, 80% power and 5% type 1 error according to the t test) is planned to be included in the study.

Hypothesis 10: : There is no difference in pain scores before, during and after suturing procedure in children watching videos with virtual reality glasses compared to the control group.

Hypothesis 11: There is a difference in pain scores before, during and after suturing in children watching videos with virtual reality glasses compared to the control group.

Hypothesis 20: There is no difference between the fear scores of children watching videos with virtual reality glasses before, during and after suturing compared to the control group.

Hypothesis 22: There is a difference between the fear scores of children watching videos with virtual reality glasses before, during and after suturing compared to the control group.

84 children will be assigned as study (42) and control (42) by block randomization method. In the study, block randomization will be done to eliminate selection bias and to provide balance in the number of individuals. The determined blocks will be created by the statistician with the codes obtained from the permutation-based computer program (https://www.randomizer.org). Then, it will be determined whether A and B are the experimental or control group by drawing lots. After the patient is evaluated according to the inclusion/exclusion criteria, self-tests will be performed by obtaining consent. In the research, single blinding will be done so that the participants will not know that they are in the experimental and control groups. In the collection of data; It is planned to use the Child Information Form, Wong-Baker Pain Scale, Child Fear Scale, which was created as a result of the literature review. In the research, video surveillance with virtual reality glasses will form the intervention group. Three minutes before watching the video with the Virtual Reality Glasses, the cartoon chosen by the child (Puzzle Tower and Z Team from the cartoons broadcast on TRT children) will be started to be watched. Pain and fear scores will be recorded before, during and after the procedure. Each child will be shown 1 episode of cartoons. This time is approximately 15 minutes. The data will be recorded before, during and after the procedure by the parent and the researcher. Researchers will definitely not perform suturing. The same health personnel will perform the suturing procedure. During the suturing procedure, data will be collected from the child by the researcher. A statistical package program will be used in the evaluation of the data. The scale mean scores of the groups will be evaluated with descriptive statistics (mean, percentage, frequency, etc.). The relevant statistics will be made according to the normality of the distribution.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7-12 years,
* Suture the emergency room on 01 October 2022 - 31 March 2023 children applying for expulsion,
* Informed volunteer signers (child and parent),
* Children without mental and developmental retardation,
* No history of epilepsy,
* Have not taken painkillers in the last 6 hours,
* There will be no stitches around the eyes and head (where the virtual reality glasses will coincide) kids
* They are children who can speak and communicate in Turkish.

Exclusion Criteria:

* Children under 7 years old and over 12 years old,
* Children who applied to the emergency room for suturing except between 01 October 2022 - 31 March 2023,
* Those who did not sign the informed consent form (child and parent),
* Children with mental and developmental retardation, with a history of epilepsy,
* Have taken painkillers in the last 6 hours,
* Stitches will be placed around the eyes and head (where the virtual reality glasses will coincide) kids
* These are children who cannot speak Turkish and cannot be communicated.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Wong Baker Pain score of the intervention group before the suture procedure | Wong Baker pain score of the intervention group three minutes before the suture procedure
  Wong Baker Pain Score; The pain level of the faces on the scale is explained to the child: "0=no pain……..10=unbearably severe pain".According to the scoring; 0-4 means mild pain, 5-6 moderate, 7-8 severe, 9-10 unbearable pain.
Wong Baker Pain Score during suture procedure of the intervention group | Wong Baker Pain Score at the time of suturing of the intervention group
  Wong Baker Pain Score; The pain level of the faces on the scale is explained to the child: "0=no pain……..10=unbearably severe pain".According to the scoring; 0-4 means mild pain, 5-6 moderate, 7-8 severe, 9-10 unbearable pain.
Wong Baker Pain Score of the control group before suture procedure | Wong Baker Pain Score of the control group three minutes before the suture procedure
  Wong Baker Pain Score; The pain level of the faces on the scale is explained to the child: "0=no pain……..10=unbearably severe pain".According to the scoring; 0-4 means mild pain, 5-6 moderate, 7-8 severe, 9-10 unbearable pain.
Wong Baker Pain Score during suture procedure of the control group | Wong Baker Pain Score at the time of suturing of the control group
  Wong Baker Pain Score;The pain level of the faces on the scale is explained to the child: "0=no pain……..10=unbearably severe pain".According to the scoring; 0-4 means mild pain, 5-6 moderate, 7-8 severe, 9-10 unbearable pain.
Child Fear Scale Score before the suture procedure of the intervention group | Child Fear Scale Score 3 minutes before suture of the intervention group
  Child Fear Scale Score; It consists of five drawn facial expressions ranging from a neutral expression (0=no anxiety) to a frightened face (4=severe anxiety) with scores ranging from 0-4.
Child Fear Scale Score during the suture procedure of the intervention group | Child Fear Score at the time of suturing of the intervention group
  Child Fear Scale Score; It consists of five drawn facial expressions ranging from a neutral expression (0=no anxiety) to a frightened face (4=severe anxiety) with scores ranging from 0-4.
Child Fear Scale Score before the suture procedure of the control group | Child Fear Scale Score 3 minutes before suture of the control group
  Child Fear Scale Score; It consists of five drawn facial expressions ranging from a neutral expression (0=no anxiety) to a frightened face (4=severe anxiety) with scores ranging from 0-4.
Child Fear Scale Score during the suture procedure of the control group | Child Fear Score at the time of suturing of the control group
  Child Fear Scale Score;It consists of five drawn facial expressions ranging from a neutral expression (0=no anxiety) to a frightened face (4=severe anxiety) with scores ranging from 0-4.
Wong Baker Pain score of the intervention group after the suture procedure | Wong Baker pain score of the intervention group three minutes after the suture procedure
  Wong Baker Pain ScoreThe pain level of the faces on the scale is explained to the child: "0=no pain……..10=unbearably severe pain".According to the scoring; 0-4 means mild pain, 5-6 moderate, 7-8 severe, 9-10 unbearable pain.;
Wong Baker Pain Score of the control group after suture procedure | Wong Baker pain score of the control group three minutes after the suture procedure
  Wong Baker Pain Score; The pain level of the faces on the scale is explained to the child: "0=no pain……..10=unbearably severe pain".According to the scoring; 0-4 means mild pain, 5-6 moderate, 7-8 severe, 9-10 unbearable pain.
Child Fear Scale Score of the intervention group after the suture procedure | Child Fear Scale Score of the intervention group three minutes after the suture procedure
  Child Fear Scale Score;It consists of five drawn facial expressions ranging from a neutral expression (0=no anxiety) to a frightened face (4=severe anxiety) with scores ranging from 0-4.
Child Fear Scale Score of the control group after the suture procedure | Child Fear Scale Score of the control group three minutes after the suture procedure
  Child Fear Scale Score;It consists of five drawn facial expressions ranging from a neutral expression (0=no anxiety) to a frightened face (4=severe anxiety) with scores ranging from 0-4.

CONTACTS AND LOCATIONS:
Overall Officials: Hacer Çetin, Study Director — Mersin University
Locations (1):
- Mersin Toros Public Hospital, Mersin, Akdeniz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Artuvan Z, Cetin H, Turkmen AS. The effect of watching videos with virtual reality glasses on pain and fear in children who undergoing suturing in the emergency department: A randomized controlled trial. J Pediatr Nurs. 2025 May-Jun;82:31-37. doi: 10.1016/j.pedn.2025.02.017. Epub 2025 Feb 28. PMID 40022763